CLINICAL TRIAL: NCT06855589
Title: Phase III Study of Hypofractionated, Dose Escalation Radiotherapy and Brachytherapy for Intermediate-risk Adenocarcinoma of the Prostate with 6 Versus 12 Months of Hormonal Manipulation
Brief Title: Optimal Duration of Hormonal Therapy for Unfavorable Intermediate-risk Prostate Cancer Patients: 6 Versus 12 Months.
Acronym: PCS-XII
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Charles LeMoyne Hospital (Other)
Responsible Party: Principal Investigator, Georges Wakil, Radiation Oncologist, MDCM, FRCPC, Principal Investigator, Clinical teaching professor, CR-CSSS Champlain-Charles-Le Moyne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCS-XII
Record Dates: First submitted 2025-02-11; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: prostate cancer; hormone therapy; stereotactic radiation therapy; brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — luprolide acetate gel depot; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 6 months of hormone therapy (Active Comparator): Patients will receive a total of two 3-month injections of a LHRH agonist
- 12 months of hormone therapy (Experimental): Patients will receive a total of four 3-month injections of a LHRH agonist
  Interventions: Drug: 12 months of Eligard; Radiation: prostate SBRT or prostate brachytherapy with radiation therapy

INTERVENTIONS:
Drug: 6 months of Eligard — Total of two 3-month injections of a LHRH agonist for total duration of 6 months
Drug: 12 months of Eligard — Total of four 3-month injections of a LHRH agonist for total duration of 12 months
  Arms: 12 months of hormone therapy
Radiation: prostate SBRT or prostate brachytherapy with radiation therapy — Patients may receive prostate stereotactic body radiation therapy or a combination of high-dose rate brachytherapy with radiation therapy; as per the treating physician's preference
  Arms: 12 months of hormone therapy

SUMMARY:
Patients with unfavorable intermediate-risk prostate cancer will be randomized between 6 versus 12 months of hormone therapy with radiation therapy. Patients may choose to receive hypofractionated radiation therapy or hypofractionated radiation therapy with high-dose rate brachytherapy. Hypofractionated radiation therapy refers to radiation therapy given fewer treatments, however higher doses per treatment.

DETAILED DESCRIPTION:
A total of 400 patients with unfavorable intermediate-risk prostate cancer will be randomized into 2 arms: The first arm will receive the standard 6-month duration of hormone therapy with concomitant radiation therapy. The second arm will receive 12 months with concomitant radiation therapy. Radiation treatment will consist of either concomitant prostate SBRT to a dose of 40 Gy/5fractions over 2 weeks or a combination of external beam radiotherapy dose of 25 Gy in 5 fractions with a high-dose rate brachytherapy boost of 15 Gy. The choice of radiation treatment will be to the investigator's discretion..Patients will be stratified according to the number of intermediate-risk factors and according to the radiation therapy type.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed adenocarcinoma of the prostate diagnosed within 6 months prior to randomization, (if longer than 6 months, needs to be approved by the central Principal Investigator).

  2. Patient has been classified as unfavorable intermediate risk as defined by one or more of the following criteria :
  * ≥ 2 of the following:
* CT2b-cT2c
* Gleason score 7 (3+4) or (4+3)
* PSA 10-20 ng/mL

  * Gleason Score 7 (4+3)
  * ≥ 50% biopsy cores positive

    3. Imaging, including CT scan and bone scan (with radiographs of suspicious areas) must be performed within 120 days prior to randomization and be negative for metastases. For patients who have started androgen suppression prior to randomization, bone scan may be done up to and including 28 days after the initiation of therapy.

    4. Pelvic and para-aortic lymph nodes must be negative on CT scan or MRI of the abdomen and pelvis performed within 120 days prior to randomization. For patients who have started androgen suppression prior to randomization, CT or MRI may be done after the start of therapy, provided it is done no more than 28 days following the start of androgen suppression therapy.

Any lymph node appearing > 1.5 cm on CT or MRI must be histologically negative by either needle aspiration or lymph node dissection performed within 12 weeks prior to randomization.

5. Patients will have had a PSA test done around the time of diagnosis. This PSA test could be repeated within 28 days prior to randomization. The PSA value used to confirm unfavorable intermediate risk disease and the value to be entered on the eligibility checklist must be the higher of these two values. These criteria will be the same regardless of whether the patient has initiated hormone therapy prior to randomization.

6. The patient may have received prior androgen suppression therapy provided that androgen suppression therapy started no more than 28 days prior to randomization.

7. The patient must not have received any cytotoxic anti-cancer therapy for prostate cancer prior to randomization. Patients may have received treatment with a 5-alpha-reductase inhibitor (e.g. Finasteride) for benign prostate hyperplasia (BPH), but must discontinue its use prior to randomization.

8. ECOG performance status must be 0 or 1. 9. Hematology and biochemistry laboratory requirements must have been done within 28-42 days prior to randomization:

1. Hemoglobin > 100 g/L
2. Absolute Neutrophils > 1.5 x 109/L
3. Platelets > 100 x 109/L
4. Serum creatinine < 1.5 x ULN 10. As it is unknown whether these treatments may affect an unborn child, adequate birth control measures should be used by the participant or his sexual partner(s) (if of reproductive potential while participating in this study).

   11. Patient consent must be obtained according to local institutional and/or University Human Experimentation Committee requirements. It will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing that such clearance has been obtained, before the trial can commence in that centre.

   12. Patients must be available for treatment and follow-ups. Investigators must ensure that the patients admitted on to this trial will be available for complete documentation of the treatment, adverse events, and follow-up visits.

   13. Prostate size must be ≤ 75 cc.

   Exclusion Criteria:
   * 1. Patients with a history of other malignancies, except: non-melanoma skin cancer; or other solid tumours curatively treated with no evidence of disease for > 5 years.

     2. The presence of small-cell or transitional-cell carcinoma in the biopsy specimen.

     3. Patients who received previous chemotherapy for carcinoma of the prostate. 4. Patients who had prior surgical treatment for carcinoma of the prostate apart from trans-urethral resection, including bilateral orchiectomy.

     5. Patients with any contraindication to pelvic radiotherapy including, but not limited to, previous pelvic radiotherapy, inflammatory bowel disease (at the discretion of the treating oncologist) or severe bladder irritability.

     6. Patients with serious non-malignant disease resulting in a life expectancy of less than 3 years.

     7. Other serious illnesses, psychiatric or medical conditions that would not permit the patient to be managed according to the protocol including active uncontrolled infection and significant cardiac dysfunction. Patients with medical conditions that would contraindicate the treatment regimen outlined in the protocol [e.g. intake of study drugs] would also NOT be eligible for the study.

     8. Known hypersensitivity to any protocol-indicated study medications. 9. Presence of bilateral hip replacement prostheses. 10. Patients with a history of severe congestive heart failure will not be eligible.

   Patients with congenital long QT syndrome or patients taking Class IA, Class III or Class IC anti-arrhythmic medications will require a cardiologist's evaluation prior to eligibility assessment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — patient must have a prostate
Enrollment: 400 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2033-03 (Estimated); Study Completion 2034-03 (Estimated)

PRIMARY OUTCOMES:
biochemical progression-free survival | 5 years
  rate of survival without a biochemical relapse. The definition of biochemical relapse is the PSA nadir + 2. The rates of biochemical relapse will be compared between the patients receiving 6 months vs 12 months of hormonal therapy.

SECONDARY OUTCOMES:
overall survival | 5 years
  rate of survival (death due to any cause)
biochemical progression-free survival | 5 years
  rate of survival without a biochemical relapse. The definition of biochemical relapse is the PSA nadir + 2. The rates of biochemical relapse will be compared between patients receiving stereotactic body radiation therapy (SBRT) vs hypofractionated radiation therapy with high-dose rate brachytherapy.
disease-specific survival | 5 years
  compare death rates due to prostate cancer between patients that received 6 months of hormone therapy versus those that received 12 months of hormone therapy.
CTCAE version 5 acute and late toxicity | 5 years
  Acute and delayed toxicity differences measured by CTCAE version 5, at or before 90 days for the acute and 90-180 days and after for the delayed toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Georges Wakil, MDCM, FRCPC, DABR, Principal Investigator — Hopital Charles Lemoyne; Tamim Niazi, MDCM, FRCPC, Principal Investigator — Jewish General Hospital
Locations (5):
- Canada (5):
  - Hôpital de Gatineau, Gatineau, Quebec
  - Hôpital Charles LeMoyne, Longueuil, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No